CLINICAL TRIAL: NCT06587919
Title: Improving Dysregulated Neural Networks With EEG-neurofeedback - A Randomized Placebo-Controlled Study
Brief Title: Improving Dysregulated Neural Networks With EEG-neurofeedback
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Imaging future (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 93533245
Record Dates: First submitted 2024-08-29; First posted 2024-09-19 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Chronic Pain; Ptsd
Keywords: EEG; neurofeedback; pain; ptsd
MeSH Terms: conditions — Chronic Pain; Stress Disorders, Post-Traumatic; Pain | interventions — Neurofeedback

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Real EEG-NF (Active Comparator): 10 EEG based neurofeedback sessions modulating the activity of the default mode network.
  Interventions: Device: Neurofeedback
- Sham EEG-NF (Sham Comparator): 10 sessions of neurofeedback another person's EEG.
  Interventions: Device: Neurofeedback

INTERVENTIONS:
Device: Neurofeedback — EEG-based neurofeedback, administered with the Neuroguide software.

SUMMARY:
Comorbid PTSD in the context of chronic pain rehabilitation is a major problem. The lack of effective and efficient methods that can be integrated into current practice is needed. The current recommended treatments for PTSD leave room for supplementary approaches to achieve symptom reduction. PTSD is characterized by specific alterations of neural activity, and the DMN is known to be involved in this. Neurofeedback is the most current approach to altering neural activity patterns towards a norm pattern found in healthy subjects.

The aim of the present study is to assess whether EEG neurofeedback compared to an active control group receiving EEG sham neurofeedback is effective in alleviating PTSD symptoms and pain intensity in patients with chronic pain and comorbid PTSD after MVCs.

DETAILED DESCRIPTION:
Prevalence and current treatment of PTSD PTSD is a debilitating mental health disorder arising from exposure to traumatic events such as war, motor vehicle accidents, crimes, and other events, threatening the lives of oneself or others involved.

The current recommended treatments for PTSD victims consist of psychotherapies and pharmacological interventions. Although 60% of PTSD patients experience improvements from a variety of trauma-focused cognitive behavior therapies, and pharmacotherapies, as many as 40% of PTSD patients do not experience symptom relief from existent therapies. Thus, the development of novel treatment alternatives is needed.

Injuries related to motor vehicle crashes (MVC) are one of the major causes of morbidity and mortality in the Western world. While physical injury and pain are the primary symptoms after MVC, between 20-40% also experience severe posttraumatic stress disorder symptoms. What is less known is that psychological distress is higher among those who have sustained a minor injury, such as whiplash injury, compared to more severe injuries, such as spinal cord injury. In particular PTSD symptoms such as hyperarousal are common after MVCs and an important mechanism in the development of chronic pain and disability after MVCs. With the mutual maintenance theory, it is suggested that pain and PTSD are mutually maintaining conditions. Indeed, PTSD is highly prevalent in the context of chronic pain rehabilitation of victims of MVCs with about 20% experiencing severe PTSD symptoms. Those with high levels of PTSD symptoms are known to experience higher levels of pain, disability, and distress. Unfortunately, targeting PTSD in pain rehabilitation is uncommon and the few existing trials that have tried to target comorbid PTSD and pain have not been sufficiently effective in alleviating pain and PTSD symptoms. Treatment resistance may be due to dysregulated brain networks that are not sufficiently targeted with traditional psychotherapeutic approaches.

A novel and promising method to target PTSD is source-localized EEG neurofeedback in that this method targets specific neural regions; thus, the treatment can be tailored to the individual patient's symptoms. As the treatment is entirely noninvasive and low-cost, the potential and the feasibility that the neurofeedback method can be employed broadly and that patients can train in between treatment sessions is considerable.

Here, we propose an investigation of the potential of standardized weighted Low-Resolution Tomography EEG neurofeedback training in treatment of comorbid PTSD in chronic pain. Our proposed study investigates the neural mechanisms hypothesized to be involved in neurofeedback training for PTSD patients. By testing, if such training can alter activity in specific target neural regions related to PTSD symptoms in our patient group, the goal is to evaluate the technique as a supplement to current therapies. We compare the active EEG neurofeedback treatment with a placebo control condition receiving sham EEG neurofeedback.

Neurofeedback In its most basic form, neurofeedback is a non-invasive technique, in which a person is trained to regulate his/her own neural activity. For psychological symptoms which are linked to dysregulated neural activity, neurofeedback may offer symptom alleviation by teaching patients to regulate relevant activity patterns themselves. By rewarding the person whenever the neural activity changes in a desired direction, the activity can be regulated or modulated. The pivotal mechanism is thus operant conditioning: A desired change in neural activity is followed by a rewarding stimulus as positive reinforcement. This reward may be appetitive to the patient, or, the reward may be in the form of a signal notifying that the training criterion is met, which in itself may be rewarding for a patient seeking symptom alleviation.

Since the 1990s, a number of studies have reported positive treatment outcomes for neurofeedback in psychiatric disorders establishing the value of neurofeedback interventions within mainstream psychiatry. Our proposed study aims at systematically registering the mechanisms involved in neurofeedback when applied to patients with comorbid PTSD and chronic pain. By doing so, we aim at furthering our understanding of the neural structures involved in posttraumatic stress symptoms and chronic pain and how neurofeedback may alter their activity patterns. This knowledge will enable the design of a specific and optimized neurofeedback training protocol for patients with PTSD and chronic pain after MVCs.

In recent decades, large-scale studies of EEG in healthy subjects across all ages and genders have been conducted to create knowledge on the characteristics of the human EEG. Such data have been processed and stored in databases making a wide range of EEG parameters available as norm data. EEG in a patient can thus be analyzed in terms of deviations from such norms. Deviations along some EEG parameters, which may be hypothesized to be involved in the targeted symptoms, can then be trained via neurofeedback to achieve greater congruence with relevant EEG parameters in healthy subjects.

Traditional neurofeedback uses one or two electrodes on the head to increase or decrease activity within a particular frequency band. Standardized Weighted Low Resolution Electromagnetic Tomography (swLORETA) is a mathematical technique to analyze the three-dimensional distribution of intracortical brain electrical activity based on surface EEG recordings. The computation enables imaging of real-time brainwave activity with a spatial resolution of less than one cubic centimeter as it divides the brain into over 12,000 voxels or pieces; this provides localization similar to that of fMRI while preserving the faster temporal resolutions of EEG. Thus, while traditional neurofeedback protocols typically utilize one or two electrode sites to train diffuse brainwave frequencies near the outer surface of the brain, source localized NF can more directly target specific brain regions even deeper within the cortex. It can also target multiple Brodmann areas simultaneously as well as give feedback on connectivity or communication between different neural sources (coherence and phase relations), enabling the option to train specific neural networks.

In combination, state-of-the-art neurofeedback offers training in deviating neural activity towards a norm mean recorded in healthy subjects, specifically targeting anatomical regions involved in symptoms.

Altered neurocircuitry in PTSD Due to the nature of the diagnostic criteria, PTSD is a heterogeneous disorder with symptom levels varying across symptom clusters. However, a key observation is changes in hyperarousal as well as self-referential processing, which refers to information relevant to oneself and is an essential component in cognitive processing. Furthermore, PTSD patients may report changes in somatic self-reference and self-perception.

In recent years, neuroscientific research has shown that many psychiatric disorders can be understood as disturbances within, or, in the relation between three basic, large brain networks. The default mode network (DMN), the salience network (SN), and the central executive networks (CEN) are concerned with self-referential processing, with external, task-related processing and with executive functions respectively. Changes in the functioning or connectivity within one network propagate to the remaining two.

Symptoms of disturbed self-referential processing in PTSD have been linked to changes in DMN connectivity. Changes in DMN may further be accompanied by an increase in SN activity, resulting in hyperarousal/heightened threat perception, and a decrease in CEN activity. Recently, PTSD symptomatology has been shown to be predicted by the level of DMN disturbance. Alterations in DMN activity and connectivity are thus strong candidates for neural correlates to altered self-referential processing in PTSD and the symptoms associated with this. Based on this knowledge, a restoration of normal activity in the DMN through neurofeedback has been suggested as a viable supplement to current treatments.

Alterations in DMN activity have also been found in acute and chronic pain states, which may reflect underlying alterations in attentional processes associated with the presence of pain itself as it has been reported that chronic pain patients also display significant attention and mental flexibility deficits. In fact, multiple studies have reported significant changes in DMN function in many chronic pain conditions. It has been suggested that the strength of the functional connections between brain regions within the DMN in chronic pain subjects relates to pain rumination, which is a measure of an individual's continuous focus on pain and its potential negative outcomes.

ELIGIBILITY:
Inclusion Criteria:

* has finished treatment at Smertecenter Syd.
* is still experiencing pain of more than 4 on the Numeric Ranking Scale (NRS).
* has been exposed to an adverse event that causes continued arousal according to the International Trauma Questionnaire.

Exclusion Criteria:

* Participants with known neurological disorders will be excluded from participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2024-09-23 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Pain intensity rating | Before every nf-session and six months after the last session.
  Average pain intensity during the last day and current pain intensity before beginning the neurofeedback session, will be assessed on an 11-point numeric rating scale (NRS) ranging from 0 (no pain) to 10 (worst imaginable pain)
EEG-power in alpha band | Before the first nf-session and after the last session (roughly six weeks later)
  37-channel EEG will be recorded, the alpha power seems to indicate cortical activity.

SECONDARY OUTCOMES:
General QoL | Assessed before first nf-session, after five weeks and after seven months.
  World Health Organization Quality of Life (WHOQOL)-Brief contains questions about how the subject feels in their everyday life, most answers are given on a five-point scale with 1 being worst/least and 5 being best/most.

CONTACTS AND LOCATIONS:
Overall Officials: Tonny Elmose Andersen, PhD, Principal Investigator — Professor at Institute of Psychology, SDU
Locations (1):
- University of Southern Denmark, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sterling M, Hendrikz J, Kenardy J, Kristjansson E, Dumas JP, Niere K, Cote J, deSerres S, Rivest K, Jull G. Assessment and validation of prognostic models for poor functional recovery 12 months after whiplash injury: a multicentre inception cohort study. Pain. 2012 Aug;153(8):1727-1734. doi: 10.1016/j.pain.2012.05.004. Epub 2012 Jun 1. PMID 22658881
- [Background] Siqveland J, Hussain A, Lindstrom JC, Ruud T, Hauff E. Prevalence of Posttraumatic Stress Disorder in Persons with Chronic Pain: A Meta-analysis. Front Psychiatry. 2017 Sep 14;8:164. doi: 10.3389/fpsyt.2017.00164. eCollection 2017. PMID 28959216
- [Background] Sharp TJ, Harvey AG. Chronic pain and posttraumatic stress disorder: mutual maintenance? Clin Psychol Rev. 2001 Aug;21(6):857-77. doi: 10.1016/s0272-7358(00)00071-4. PMID 11497210
- [Background] Ravn SL, Hartvigsen J, Hansen M, Sterling M, Andersen TE. Do post-traumatic pain and post-traumatic stress symptomatology mutually maintain each other? A systematic review of cross-lagged studies. Pain. 2018 Nov;159(11):2159-2169. doi: 10.1097/j.pain.0000000000001331. PMID 29994992
- [Background] Ipser J, Seedat S, Stein DJ. Pharmacotherapy for post-traumatic stress disorder - a systematic review and meta-analysis. S Afr Med J. 2006 Oct;96(10):1088-96. PMID 17164942
- [Background] Craig A, Tran Y, Guest R, Gopinath B, Jagnoor J, Bryant RA, Collie A, Tate R, Kenardy J, Middleton JW, Cameron I. Psychological impact of injuries sustained in motor vehicle crashes: systematic review and meta-analysis. BMJ Open. 2016 Sep 8;6(9):e011993. doi: 10.1136/bmjopen-2016-011993. PMID 27609849
- [Background] Buitenhuis J, de Jong PJ, Jaspers JP, Groothoff JW. Relationship between posttraumatic stress disorder symptoms and the course of whiplash complaints. J Psychosom Res. 2006 Nov;61(5):681-9. doi: 10.1016/j.jpsychores.2006.07.008. PMID 17084147
- [Background] Bradley R, Greene J, Russ E, Dutra L, Westen D. A multidimensional meta-analysis of psychotherapy for PTSD. Am J Psychiatry. 2005 Feb;162(2):214-27. doi: 10.1176/appi.ajp.162.2.214. PMID 15677582
- [Background] Andersen TE, Ravn SL, Armfield N, Maujean A, Requena SS, Sterling M. Trauma-focused cognitive behavioural therapy and exercise for chronic whiplash with comorbid posttraumatic stress disorder: a randomised controlled trial. Pain. 2021 Apr 1;162(4):1221-1232. doi: 10.1097/j.pain.0000000000002117. PMID 33086286
- [Background] Andersen TE, Lahav Y, Ellegaard H, Manniche C. A randomized controlled trial of brief Somatic Experiencing for chronic low back pain and comorbid post-traumatic stress disorder symptoms. Eur J Psychotraumatol. 2017 May 30;8(1):1331108. doi: 10.1080/20008198.2017.1331108. eCollection 2017. PMID 28680540
- [Background] Andersen TE, Ellegaard H, Schiottz-Christensen B, Mejldal A, Manniche C. Somatic Experiencing(R) for patients with low back pain and comorbid posttraumatic stress symptoms - a randomised controlled trial. Eur J Psychotraumatol. 2020 Aug 18;11(1):1797306. doi: 10.1080/20008198.2020.1797306. PMID 33029333